CLINICAL TRIAL: NCT07101653
Title: From Muscle to Brain: Exercise Induces Structural Brain Changes, Irisin Elevation, and Functional Recovery in Multiple Sclerosis - Exploring the Interrelationships
Brief Title: Exercise-Induced Irisin and Brain Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan Bilek, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/13-37
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Irisin; Brain Volume
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This single-blind, randomized controlled trial
Who Masked: Investigator
Masking Description: All clinical assessments will be performed by a blinded neurologist to eliminate measurement bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Based on current recommendations for individuals with MS, the PRT program will last 12 weeks and will include three sessions per week, each lasting 60-90 minutes at 60-80% of one-repetition maximum.
  Interventions: Other: Exercise
- No intervantion (No Intervention): No intervantion

INTERVENTIONS:
Other: Exercise — According to current clinical guidelines for multiple sclerosis patients, the progressive resistance training (PRT) protocol will be implemented as follows: a 12-week intervention consisting of three supervised 60-90 minute sessions per week at 60-80% of one-repetition maximum intensity. All training sessions will be conducted under the direct supervision of a certified physiotherapist to ensure proper technique adherence and safety throughout the intervention period
  Arms: Exercise

SUMMARY:
This single-blind, randomized controlled trial will employ a two-arm parallel design (exercise group vs. control group) with a 12-week intervention period. Sex-stratified randomization will be implemented using SPSS 25.0 (IBM Corporation, Armonk, NY, USA) to ensure balanced group allocation. All outcome measures will be assessed at baseline and post-intervention.

DETAILED DESCRIPTION:
The exercise intervention will consist of supervised progressive resistance training sessions conducted three times weekly (with a minimum 48-hour rest period between sessions) at Firat University Hospital. Control participants will maintain their usual daily activities without participating in any structured exercise programs.

A blinded neurologist will perform all clinical assessments to eliminate measurement bias. To control for circadian variations, all evaluations will be scheduled at consistent times of day for each participant. Environmental conditions will be strictly maintained during testing sessions (ambient temperature: 21-22°C; humidity: 55-60%).

This study will be designed and reported in accordance with CONSORT guidelines for randomized trials, incorporating all essential elements for transparent randomized controlled reporting, including allocation concealment, blinding procedures, and intention-to-treat principles.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed relapsing-remitting multiple sclerosis (RRMS) diagnosis according to revised McDonald criteria (2017)
* Aged 19-65 years (inclusive)
* Mild-to-moderate disability (EDSS score 1.0-5.5)
* No corticosteroid treatment within the previous 3 months

Exclusion Criteria:

* Acute MS relapse within 90 days prior to enrollment
* Regular participation in structured exercise programs (>3 hours/week)
* Comorbid conditions that may limit exercise participation, including; significant orthopedic impairments, unstable cardiopulmonary conditions and other systemic disorders affecting physical activity
* Standard MRI contraindications (metallic implants, claustrophobia, etc.)
* Concurrent neurological disorders (other than MS)
* Initiation or modification of disease-modifying therapy within 6 months
* Severe spasticity (Modified Ashworth Scale ≥3 in any major muscle group)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
MRI Acquisition and Volumetric Analysis | 12 weeks
  Volumetric brain analysis will be conducted using VolBrain, an open-access automated segmentation platform for brain MRI.
Serum irisin hormone measurement | 12 weeks
  All patients will be asked to provide blood samples in the morning following their overnight (12 h) fast before and after the study. The unit pg/ml will be used for serum irisin.

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composite | 12 weeks
  Multiple Sclerosis Functional Composite (MSFC) is a standardized, quantitative tool used to assess disability and functional changes in individuals with multiple sclerosis (MS).

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I dont want to share IPD with other researchers